CLINICAL TRIAL: NCT02324881
Title: A Pilot Study for a Pain Management Smartphone Application for Patients Undergoing Radiation Therapy for Locally Advanced Head and Neck Cancer
Brief Title: Pain Management Smartphone Application for Patients With Stage III-IV Head and Neck Cancer Undergoing Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Friedman, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VICC HN 14122; NCI-2014-02426 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICCHN14122 (Other: Vanderbilt-Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Head and Neck Cancer; Pain; Lung Cancer; Esophageal Cancer
Keywords: smartphone; application; pain management
MeSH Terms: conditions — Head and Neck Neoplasms; Pain; Lung Neoplasms; Esophageal Neoplasms; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health Services Research (PMSA) (Experimental): Patients/caregivers are instructed to download the PMSA and are demonstrated how to properly use the application. Beginning on the first day of radiation therapy (day 1), patients are instructed to use the PMSA for the duration of their radiation therapy (up to day 50). The patient will fill out a satisfaction questionnaire at the completion of their treatment (Questionnaire administration). The timing of use may change depending on the availability of the app. The use of the app is classified as the "telephone-based intervention" per NCI.
  Interventions: Behavioral: Telephone-Based Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Telephone-Based Intervention — Use PSMA
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies a pain management smartphone application for monitoring pain in patients with locally advanced head and neck cancer who are undergoing radiation therapy. The study is also open to patients with esophageal or lung cancer. A smartphone application may allow patients to assess their symptoms in a manner that is closer to real-time than having to recall pain episodes during once weekly on-treatment visits with a health care provider. This real-time monitoring may improve the timing and efficacy of interventions leading to better pain-control and quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Obtain consumer input to determine the optimal way to address and monitor the patient's symptoms.

II. Train patients to use the pain management smartphone application (PMSA) and determine the compliance characteristics and the number of additional on-treatment visits (OTVs) prompted by usage of the application.

OUTLINE:

Selected patients are interviewed for input that will help guide the wording of questions of the PMSA. All patients/caregivers are then instructed to download the PMSA and are demonstrated how to properly use the application. Beginning on the first day of radiation therapy (day 1), patients are instructed to use the PMSA for the duration of their radiation therapy (up to day 50), although the timing may change based on the availability of the app.

ELIGIBILITY:
Inclusion Criteria:

* Radiation oncology patients undergoing 5-7 weeks of definitive radiation therapy for head and neck, esophageal or lung cancer.
* Ability to understand and the willingness to use the PMSA on the patient's personal smartphone
* Displays ability to use and understand the PMSA as evidenced by successful response to alarm and successful entries while monitored by the principal investigator (PI)
* Willing and able to provide informed consent and fill out demographic, disease, and pain assessment questionnaires
* English speaking

Exclusion Criteria:

* Radiation oncology patients undergoing palliative courses of radiation
* Patients who do not own smartphones
* Patients who are unable to successfully respond to the PMSA alarm and properly enter their data
* Patients who are unable to eat and drink normally
* Patients who are unable to validate their understanding of the pain scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Compliance characteristics of patients' use of the pain management smartphone application | Up to day 50
  Summaries of feasibility will be generated using rates (percentages). Descriptive statistics will be used to summarize patient ratings of satisfaction regarding the PMSA, instruction, usage, and future recommendation.

SECONDARY OUTCOMES:
Number of additional OTVs prompted by usage of the application | Up to day 50
  The additional OTVs per patient will analyzed with descriptive statistics, such as frequency distributions, means, medians and measures of variability will be used to describe the OTV number changes.

OTHER OUTCOMES:
Ability to obtain consumer input to determine the optimal way to address and monitor the patient's symptoms | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Friedman, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/